CLINICAL TRIAL: NCT00667108
Title: A Randomized, Double-Blind, Single-Dose, Placebo-Controlled, Multicenter Study of Gabapentin 250 mg and 500 mg in Transient Insomnia Induced by a Sleep Phase Advance
Brief Title: A Study of Single-Dose Gabapentin in Transient Insomnia Induced by a Sleep Phase Advance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9451140
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2008-04

CONDITIONS: Transient Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gabapentin 250 mg (Experimental)
  Interventions: Drug: Gabapentin
- Gabapentin 500 mg (Experimental)
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 250 mg oral capsule 30 minutes prior to bedtime
  Arms: Gabapentin 250 mg
Drug: Gabapentin — Gabapentin 500 mg oral capsule 30 minutes prior to bedtime
  Arms: Gabapentin 500 mg
Drug: Placebo — Matched placebo 30 minutes prior to bedtime
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of gabapentin as compared to placebo on sleep, using subjective sleep measurements, in subjects with transient insomnia induced by a sleep phase advance.

ELIGIBILITY:
Inclusion Criteria:

* Aged >/= 18 years
* Females of child-bearing potential using medically-acceptable method of birth control >/= 1 month prior to screening

Exclusion Criteria:

* Current or recent history (within 2 years) of sleep disorder (excessive snoring, obstructive sleep apnea, chronic painful condition)
* Recreational drug use within past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 784 (Actual)
Dates: Start 2004-10; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Subjective sleep latency | Hour +8

SECONDARY OUTCOMES:
Subjective assessment of sleep refreshment | Hour +8
Subjective assessment of sleep quality | Hour +8
Karolinska Sleep Diary-Sleep (KSD) Quality Index | Hour +8
KSD individual scores | Hour +8
Digit Symbol Substitution Test | Hour +8
Buschke Selective Reminding Test (immediate recall score, long term storage score, total number of intrusions, delayed recall score) | Hour +8
Stanford Sleepiness Scale | Hour +13
Vital signs | Hour +8
Adverse events | Hour +13
Subjective number of awakenings | Hour +8
Subjective wake after sleep onset | Hour +8
Subjective total sleep time | Hour +8

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Mount Laurel, New Jersey
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Dallas, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451140&StudyName=A%20Study%20of%20Single-Dose%20Gabapentin%20in%20Transient%20Insomnia%20Induced%20by%20a%20Sleep%20Phase%20Advance